CLINICAL TRIAL: NCT00002076
Title: Pilot Study of Oral Fluconazole in the Treatment of Acute Cryptococcal Meningitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 012J; 056-162
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-02

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Fluconazole; Administration, Oral; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To evaluate the safety and effectiveness of fluconazole as treatment for acute cryptococcal meningitis in AIDS patients. Both newly diagnosed and relapsed patients are eligible.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiviral therapy such as zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.
* Aerosolized pentamidine.

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Written informed consent must be obtained for each patient, either from the patient himself or from the patient's legal guardian.

* No prior systemic antifungal therapy for cryptococcosis.
* Success of prior therapy must have been documented by negative cerebrospinal fluid (CSF) culture at the end of therapy. Following prior therapy, such patients may not have received more than 1 mg/kg/wk amphotericin B in the 4 weeks before entry into study.

Prior Medication:

Allowed:

* Antiviral therapy such as zidovudine.
* Prophylaxis for Pneumocystis carinii pneumonia.
* Aerosolized pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease defined by specified lab values.
* Patients who are unable to take oral medication.
* Unlikely to survive more than 2 weeks.
* Renal impairment.

Concurrent Medication:

Excluded:

* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications other than aerosolized pentamidine.
* Excluded within 4 weeks of study entry:
* Greater than 1 mg/kg/wk amphotericin B.
* Any exceptions to these prohibitions of concomitant medications must be approved by Pfizer Central Research.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy to or intolerance of imidazoles or azoles.
* Moderate or severe liver disease defined by specified lab values.
* Patients who are unable to take oral medication.
* Life expectancy of < 2 weeks.
* Any condition that may impair absorption of oral medication.

Prior Medication:

Excluded:

* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications other than aerosolized pentamidine.
* Excluded within 4 weeks of study entry:
* Greater than 1 mg/kg/wk amphotericin B.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Summitt Med Ctr / San Francisco Gen Hosp, Oakland, California
  - Cornell Univ Med Ctr, New York, New York
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania